CLINICAL TRIAL: NCT05569837
Title: The Effect of Irregular Meal Pattern Providing Hypo-energetic Diet on Energy Expenditure, Metabolism and Circadian Rhythm: a Randomized Controlled Trial
Brief Title: The Effect of Irregular Meal Pattern Providing Hypo-energetic Diet on Energy Expenditure and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Moira Taylor, Principal Investigator, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 473- 2001
Record Dates: First submitted 2022-09-21; First posted 2022-10-06 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Metabolic Disturbance; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular meal pattern (Experimental): Participants will follow a regular meal pattern for 14 days
  Interventions: Other: Regular meal pattern
- Irregular meal pattern (Experimental): Participants will follow an irregular meal pattern for 14 days
  Interventions: Other: Irregular meal pattern

INTERVENTIONS:
Other: Regular meal pattern — 6 meals every day
  Arms: Regular meal pattern
Other: Irregular meal pattern — It consists of consuming a different number of meals every day (between 3 and 9).
  Arms: Irregular meal pattern

SUMMARY:
In this study we will compare the effect of two different meal patterns. Firstly, participants will consume a diet providing their estimated energy requirement for a 7 day standardisation period (6 meals per day). After a one day laboratory visit, this will be followed by a 14 day intervention period when participants will randomly follow a regular meal pattern (6 meals/d) or an irregular meal pattern (3-9 meals/d). Following a further laboratory visit day, they will then consume the previous standardisation diet for a further 3 days. The energy intake provided will be calculated to provide less energy than subjects are using which may result in approximately 2kg of weight loss. Participants will attend a screening visit in which they will complete questionnaires on medical health, eating habits and physical activity. In the laboratory visit, participants will be fasting and for 3 h after intake of a test drink, measurements will be taken of energy expenditure, fasting glucose, fasting gut hormones, fasting lipids and fasting insulin. A test meal will be offered. A questionnaire of subjective appetite ratings will be assessed while fasting, after the test drink, after the test meal, and during the intervention. Continuous interstitial glucose monitoring will be undertaken during the whole study period, Core body temperature will be measured before and after the intervention period. Also, wrist temperature will be measured during the whole study period.

DETAILED DESCRIPTION:
Experimental protocol:

28 women who are a healthy weight or overweight (aged 18-45 years) will be recruited to a randomized parallel trial to follow one of two 14-d hypo-energetic diets. Firstly, participants will consume a diet providing their estimated energy requirement (6 meals/day) for a 7 day standardisation period. After a one day laboratory visit, this will be followed by a 14 day intervention period when participants will follow a regular meal pattern (6 meals/d) or an irregular meal pattern (3-9 meals/d) (energy deficit of 800kcal/ 24h in both diets) (identical foods provided on both interventions whilst otherwise free living). Following a further laboratory visit day, they will then consume the previous standardisation diet providing their estimated energy requirement (6 meals/day) for a further 3 days. All foods to be consumed during the study will be provided to free of charge. These will comprise foods commonly consumed in the British diet and will be consumed in amounts designed to provide 800kcal/24h less than estimated energy requirements in the intervention period. Participants will attend the laboratory visits fasting and a blood sample will be obtained for fasting glucose, insulin and lipids. A test drink will then be given and over the following three hours measurements will be taken of energy expenditure (TEF). An ad libitum pasta test meal will be offered three hours after the test drink has been given. Subjective appetite ratings will be assessed while fasting, after the test drink, after the ad libitum meal, and during the intervention. Continuous interstitial glucose monitoring will be undertaken throughout the study. Ambulatory activity pattern measurement will be assessed in the intervention period. Core body temperature will be measured during the last 3 days of the first standardisation period, and during the final three standardisation days. Peripheral body temperature will be measured throughout the study period using a small i- button secured to the wrist. The study will commence at the early phase of the menstrual cycle (days1-7). A constant sleep-wake (and light exposure) routine will be followed for the whole study period which will be assessed by a written questionnaire form

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30 kg/m2,
* Age between 18 and 45y,
* Non-smokers,
* Non high-alcohol consumers (≥ 14 units/week),
* Regular menstruation or on the oral contraceptive pills,
* Their weight is stable during the previous 3 months,
* No self-reported history of serious medical conditions and not under medication.

Exclusion Criteria:

* Pregnant or lactating women
* Smokers
* High-alcohol consumers (≥ 14 units/week)
* Subjects with high score for depression using Becks Depression Inventory
* subjects Eating Attitudes Test (EAT-26) score >20
* Subjects who on diet or seeking to lose weight
* Subjects with high consumption of coffee or tea > 3 cups/day

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline thermic effect of food in kcal at 2 weeks intervention | Over 3 hours for 2 days
  Indirect calorimetry (GEM system; Europa Scientific Ltd.) will be used to determine the resting energy expenditure (REE) and thermic effect of food (TEF). REE will be measured in the fasted state for 20 min. The TEF will be measured for periods of 15 min at 30-min intervals during the 3 h after test drink (milkshake) consumption.

SECONDARY OUTCOMES:
Change from baseline body Weight in kilograms at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  Body weight
Change in subjective appetite | 2 days in lab visit, 1 day pre-intervention standardization period, 1 day post-intervention standardization period and 2 days in intervention period
  a booklet will be given to record the subjective appetite (hunger, fullness and desire to eat) using visual analogue scales (VAS) before and after each single meal on:
  1. The last day of the pre-standardization period,
  2. The first day of the post-intervention period.
  3. Pre-lab visit day.
  4. Post-lab visit day.
  5. Day 7 during the intervention period.
  6. Day 14 during intervention period.
Continuous interstitial glucose | 26 days
  Continuous interstitial glucose will be undertaken using a continuous glucose monitor (CGM) the FreeStyle Libre System during the whole study period
Change from baseline fasting glucose in mmol/L at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting sample of serum glucose
Change from baseline fasting insulin in mlU/L at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting sample of serum insulin
Change from baseline fasting lipids in mmol/L at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting sample of serum total cholesterol, HDL cholesterol, LDL cholesterol and triacylglycerol.
Change from baseline fasting glucagon-like peptide1 in pM at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting plasma glucagon-like peptide1(GLP-1).
Change from baseline fasting peptide YY in pg/ml at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting plasma peptide YY (PYY).
Change from baseline fasting ghrelin in pg/ml at 2 weeks intervention | 1 day before intervention and 1 day after intervention
  A fasting blood samples will be taken, just before ingestion of the test drink to assess the mean of the fasting plasma ghrelin.
Change from baseline core body temperature in Celsius at 2 weeks intervention | 3 days in pre and post intervention
  Core temperature will be assessed using an ingestible telemetry pill and associated monitor (e-Celsius Performance pill and monitor e-Celcius™ BodyCap).
Peripheral wrist temperature in Celsius | 26 days
  Wrist temperature will be assessed through a wireless iButton data logger

CONTACTS AND LOCATIONS:
Overall Officials: Moira Taylor, PhD, Principal Investigator — University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta-analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When requested
Access Criteria: On receipt of requests, data will be made accessible if agreed by the University of Nottingham

REFERENCES:
- [Background] Alhussain MH, Macdonald IA, Taylor MA. Irregular meal-pattern effects on energy expenditure, metabolism, and appetite regulation: a randomized controlled trial in healthy normal-weight women. Am J Clin Nutr. 2016 Jul;104(1):21-32. doi: 10.3945/ajcn.115.125401. Epub 2016 Jun 15. PMID 27305952
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Regular meal frequency creates more appropriate insulin sensitivity and lipid profiles compared with irregular meal frequency in healthy lean women. Eur J Clin Nutr. 2004 Jul;58(7):1071-7. doi: 10.1038/sj.ejcn.1601935. PMID 15220950
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Decreased thermic effect of food after an irregular compared with a regular meal pattern in healthy lean women. Int J Obes Relat Metab Disord. 2004 May;28(5):653-60. doi: 10.1038/sj.ijo.0802616. PMID 15085170
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Beneficial metabolic effects of regular meal frequency on dietary thermogenesis, insulin sensitivity, and fasting lipid profiles in healthy obese women. Am J Clin Nutr. 2005 Jan;81(1):16-24. doi: 10.1093/ajcn/81.1.16. PMID 15640455